CLINICAL TRIAL: NCT05866770
Title: A Feasibility, Prospective, Multi-centre, Repeated Measures Investigation Evaluating the Application of Hearing Aid Technologies to Signal Processing for Adult Cochlear Implant Recipients
Brief Title: A Study Evaluating the Application of Hearing Aid Technologies to Signal Processing for Adult Cochlear Implant Recipients
Acronym: HATSI-MB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AI5837
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- U8 then N8 (Other): Participants in this arm receive U8 followed by N8
  Interventions: Device: U8; Device: N8 sound processor
- N8 then U8 (Other): Participants in this arm receive N8 followed by U8
  Interventions: Device: U8; Device: N8 sound processor

INTERVENTIONS:
Device: U8 — The U8 Research System
Device: N8 sound processor — Nucleus 8 sound processor

SUMMARY:
A feasibility, prospective, multi-centre, repeated measures investigation evaluating the application of hearing aid technologies to signal processing for adult cochlear implant recipients

DETAILED DESCRIPTION:
The Research System is comprised of several components: the processing unit, fitting software and accessories. The sound processor converts sounds into electrical signals, which it sends, via a coil, to an implant to provide hearing sensation. The application of hearing aid technologies to Cochlear Implant recipients may provide benefit through matching the signal processing technologies across ears for bimodal listeners, enhance performance for CI-alone listening, and potentially lead to efficiency in algorithm development.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* User of CI600, CI500 or CI24RE implant
* At least 3 months experience with a TGA approved Nucleus cochlear implant in at least one ear
* Fluent speaker of English
* A word speech recognition score of 20% or more when using the cochlear implant alone*
* Willing and able to provide written informed consent *This can be based on clinical data if collected within the last 12 months

Exclusion criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families: immediate family is defined as a spouse, parent, child, or sibling
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device. (Unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent correct monosyllabic word scores. | 3 months
  To determine whether the research system provides non-inferior performance to the Nucleus 8 sound processor for monosyllabic words in quiet CNC words at 60 dB SPL (sound pressure level)
  Word recognition is a score of the number of words correctly repeated, expressed as a percentage. Higher percentage scores indicate a better outcome.
Adaptive sentence in noise scores (AuSTIN) | 3 months
  To determine whether the research system provides non-inferior performance to the Nucleus 8 sound processor for sentences in noise.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Cochlear Melbourne, Melbourne E., melbourne
  - Cochlear Macquarie, Sydney, New South Wales
  - HEARnet Clinical Studies, Carlton, Victoria

IPD SHARING:
Plan to Share IPD: No